CLINICAL TRIAL: NCT04636216
Title: Open Trial of a Program to Support Parents of Children With Attention-deficit/Hyperactivity Disorder in Online Group Meetings
Brief Title: Open Trial of a Program to Support Parents of Children With Attention-deficit/Hyperactivity Disorder (ADHD)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Florida International University (Other)
Responsible Party: Principal Investigator, Dr. Greg Fabiano, Professor, Florida International University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB-20-0484
Record Dates: First submitted 2020-10-22; First posted 2020-11-19 (Actual); Last update posted 2021-10-28 (Actual); Status verified 2021-10

CONDITIONS: ADHD
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity

STUDY DESIGN:
Intervention Model Description: Open, single-group trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Community Parent Education Program (COPE) parent training program (Experimental): Parents will enroll in an 8-week, group parenting program.
  Interventions: Behavioral: COPE parent training

INTERVENTIONS:
Behavioral: COPE parent training — Weekly 1.5 hour parent training meetings for eight weeks

SUMMARY:
Behavioral parent training is an evidence-based treatment for ADHD. The intervention can be implemented individually, or in groups. Currently, group-based parent training programs require considerable coordination, including ascertainment of a large physical space, the coordination of all families traveling to the same location at the same time, and the require for the provision of childcare. Innovations in online connectivity and ease of implementation of online support applications (e.g., Zoom) may reduce these barriers. However, it is necessary to investigate the feasibility and promise of the online approach to ensure it supports parents effectively.

DETAILED DESCRIPTION:
This study will utilize a pre-post, open trial design as the primary aim is to investigate feasibility. Approximately sixty parents will complete prepost ratings of parenting behaviors and measures of child functioning. They will also complete post treatment measures of satisfaction and open-ended questions about feasibility and suggestions for future iterations of the approach. Process measures will include data collection related to attendance and engagement in the activities. Risks include breach of confidentiality and a lack of effectiveness of the intervention for the child's presenting problems. Benefits include the parent receiving an effective intervention.

ELIGIBILITY:
Inclusion Criteria:

* ADHD diagnosis
* Intelligence Quotient (IQ) greater than or equal to 70
* At least 1 parent/guardian who can attend zoom sessions
* Access to reliable internet connection for zoom meetings

Exclusion Criteria:

* Evidence of psychosis, suicidal behaviors, or autism level 2/3

Ages: 5 Years to 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 14 (Actual)
Dates: Start 2020-11-03 (Actual); Primary Completion 2021-05-30 (Actual); Study Completion 2021-05-30 (Actual)

PRIMARY OUTCOMES:
Observations of parenting behaviors during parent-child interaction | 8 weeks
  Dyadic Parent Child Interaction code frequency counts for the categories of Negative Talk, Praise, and Commands
Impairment Rating Scale | 8 weeks
  Average score across domains with scores ranging from 0 (No problem) to 6 (Extreme problem)

CONTACTS AND LOCATIONS:
Overall Officials: Gregory A Fabiano, Ph.D., Principal Investigator — Florida International University
Locations (1):
- Center for Children and Families, Amherst, New York, United States

IPD SHARING:
Plan to Share IPD: No